CLINICAL TRIAL: NCT04778683
Title: THE EFFECT OF VIRTUAL REALITY ON CHILDREN'S ANXIETY, FEAR, AND PAIN LEVELS BEFORE CIRCUMCISION IN TURKEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OMU-B.30.2.ODM.0.2
Record Dates: First submitted 2021-02-13; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: to Have a Circumcision Operation
Keywords: circumcision; child; virtual reality; anxiety; fear; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This randomized controlled study was conducted a pediatric hospital in Turkey for circumcision between June and September 2019. The sample size for the study was calculated using the G-Power 3.0.10 program and t-test for comparison of two independent groups with an effect size of 0.8, an alpha level and margin of error of 0.05, and a power of 95%. The sample size was determined to be 70; each of the experimental and control groups included 35 children. Data were collected from 78 children. A randomized block design method was used to randomize the participants to the groups. The randomization list was prepared by a third person and was given to the investigator only during the application.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sociodemographic data of the children and their mothers were collected using the participant information form. Then, the children rated their fear and anxiety on the scales using a pen. Similar assessments were performed by their mothers and the investigator. The investigator explained the use of VR glasses to the children in the VR group. After the surgery, the children, their mothers, and the investigator re-evaluated the fear and anxiety in children using the CFS and the CAM-S. The pain levels in children during the postoperative period were evaluated by both their mothers and the nurse. The same evaluations were performed in children in the control group who received routine clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): The investigator explained the use of VR glasses to the children in the VR group. The investigator selected two VR programs to be watched by the children. In the VR program named Amazon, the child perceives himself to be walking among the trees in the Amazon forests. The other VR program gives the child a feeling of water skiing.
  Interventions: Procedure: Virtual Reality
- Control Group (No Intervention): The same evaluations were performed in children in the control group who received routine clinical care.

INTERVENTIONS:
Procedure: Virtual Reality — The investigator explained the use of VR glasses to the children in the VR group. The investigator selected two VR programs to be watched by the children. In the VR program named Amazon, the child perceives himself to be walking among the trees in the Amazon forests. The other VR program gives the child a feeling of water skiing. Before commencement of the study, the VR applications were administered to five children aged between five and ten years, and these children shared no negative feedback about the VR programs. Before the surgery, the children were allowed to watch the VR program of their choice, the average duration of which was 4.5 minutes, using the VR glasses. Parts of the device that come in contact with the children's faces were cleaned before each application
  Arms: VR Group

SUMMARY:
Background: Circumcision is one of the most common surgical interventions in boys, and boys undergoing this procedure experience anxiety and fear during the preoperative period. In addition, postoperative pain in children is reported to be associated with anxiety and fear.

Aim: This study aimed to examine the effects of using a virtual reality (VR) application before circumcision on the pre- and postoperative anxiety and fear levels and postoperative pain symptoms in children.

Material and Methods: This randomized controlled experimental study included 5-to 10-year-old boys referred to a pediatric hospital for circumcision between June and September 2019. Randomization was performed using the randomized block design, and the subjects were divided into control (n = 38) and experimental (n = 40) groups. The data were collected using a participant information form, the children's fear scale (CFS), the children's anxiety meter scale (CAM-S), and the Wong-Baker Faces Pain Rating Scale; data were analyzed using SPSS 22.0 package program. The data were evaluated using descriptive statistics; the chi-square test was used to assess the sociodemographic data, the Mann-Whitney U test was used to compare two independent groups, the Wilcoxon T-test was used to compare intra-group preoperative and postoperative values, and the Spearman Correlation test was used to examine the relationship between anxiety, fear and pain scores.

Keywords: Circumcision, child, virtual reality, anxiety, fear, pain.

DETAILED DESCRIPTION:
This randomized controlled study was included 5-to 10-year-old boys who were referred to a pediatric hospital in Turkey for circumcision between June and September 2019. The sample size for the study was calculated using the G-Power 3.0.10 program and t-test for comparison of two independent groups with an effect size of 0.8, an alpha level and margin of error of 0.05, and a power of 95%. The sample size was determined to be 70; each of the experimental and control groups included 35 children. Data were collected from 98 children. Of them, 14 children were excluded from the study because two could not obtain approval from their families to participate in the study, four had previous surgical interventions, six had chronic and mental illnesses, and two had vision problems. The inclusion criteria for the study were agreement to participation in the study, age between 4 and 10 years, no vision or hearing problems, no history of surgical intervention, and no chronic and mental health problems. Children who met the inclusion criteria and who had written and verbal consents from their parents for participation in the study were divided into 2 groups. The experimental group consisted of 40 children who received a VR application, and the control group consisted of 38 children who received standard healthcare. A randomized block design method was used to randomize the participants to the groups. The randomization list was prepared by a third person and was given to the investigator only during the application.

Instruments The data were collected using a participant information form to obtain details about baseline characteristics; children's fear scale (CFS) and children's anxiety meter scale (CAM-S) were used to evaluate fear and anxiety in children during both the pre- and postoperative periods, and the Wong-Baker faces pain rating scale (WBS) was used to evaluate the levels of postoperative pain in children. A white colored "VR BOX 3.0" with VR glasses (a headset with a screen covering the children's eyes) was used in this study. It was compatible with iOS and Android operating systems and 4-6-inch screen smartphones. The VR device, which is activated through applications installed on smartphones, divides the image into two equal windows, providing the necessary viewfinder range for panoramic view. The distance between the mobile phone and the lens can be adjusted for each user. The VR glasses do not require any power or electrical connection, except the mobile phone, during their use. The weight of the VR glasses is 0.414 kg. Soundproof headsets are used to provide immersive VR.

Procedure Sociodemographic data of the children and their mothers were collected using the participant information form. Then, the children rated their fear and anxiety on the scales using a pen. Similar assessments were performed by their mothers and the investigator. The investigator explained the use of VR glasses to the children in the VR group. The investigator selected two VR programs to be watched by the children. In the VR program named Amazon, the child perceives himself to be walking among the trees in the Amazon forests. The other VR program gives the child a feeling of water skiing. Before commencement of the study, the VR applications were administered to five children aged between five and ten years, and these children shared no negative feedback about the VR programs. Before the surgery, the children were allowed to watch the VR program of their choice, the average duration of which was 4.5 minutes, using the VR glasses. Parts of the device that come in contact with the children's faces were cleaned before each application. After the surgery, the children, their mothers, and the investigator re-evaluated the fear and anxiety in children using the CFS and the CAM-S. The pain levels in children during the postoperative period were evaluated by both their mothers and the nurse. The same evaluations were performed in children in the control group who received routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participation in the study,
* age between 5 and 10 years,
* no vision or hearing problems,
* no history of surgical intervention,
* no chronic and mental health problems

Exclusion Criteria:

* no agreement to participation in the study,
* age lower than 5 and upper 10 years,
* to have vision or hearing problems,
* to have history of surgical intervention,
* to have chronic and mental health problems

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate Anxiety with anxiety meter scale | VR practice one hour before circumcision
  VR practice before circumcision reduces pre-operative and post-operative anxiety level
Evaluate Fear with fear meter scale | VR practice one hour before circumcision
  VR practice before circumcision reduces pre-operative and post-operative fear level
Evaluate Pain with Wong-Baker Faces Pain Rating Scale | VR practice one hour before circumcision
  VR practice before circumcision reduces postoperative pain symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tural Büyük, Assoc. Prof., Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No